CLINICAL TRIAL: NCT01568034
Title: A Double-blind, Randomised, Placebo-controlled, Cross-over Study to Investigate the Tolerability and Effect of Three Single-dose Regimens of BIA 9-1067 on the Levodopa Pharmacokinetics, Motor Response, and Erythrocyte Soluble Catechol-O-methyltransferase Activity in Parkinson's Disease Patients Concomitantly Treated With Levodopa/Dopa-decarboxylase Inhibitor
Brief Title: A Study to Investigate the Tolerability and Effect of Three Single-dose Regimens of BIA 9-1067
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BIA-91067-201; 2008-003869-72 (EudraCT Number)
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Results first posted 2015-01-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2014-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; BIA 9-1067
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone; carbidopa, levodopa drug combination; Levodopa

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment Sequence A (Experimental): Treatment Sequence A Period 1 - 25 mg BIA 9-1067 Period 2 - 50 mg BIA 9-1067 Period 3 - 100 mg BIA 9-1067 Period 4 - Placebo
  Levodopa/Carbidopa combination were given to half of the volunteers and Levodopa/Benzerazide to the other half
  Interventions: Drug: BIA 9-1067; Drug: Placebo; Drug: Levodopa/Carbidopa; Drug: Levodopa/Benzerazide
- Treatment Sequence B (Experimental): Treatment Sequence B Period 1 - Placebo Period 2 - 25 mg BIA 9-1067 Period 3 - 50 mg BIA 9-1067 Period 4 - 100 mg BIA 9-1067
  Levodopa/Carbidopa combination were given to half of the volunteers and Levodopa/Benzerazide to the other half
  Interventions: Drug: BIA 9-1067; Drug: Placebo; Drug: Levodopa/Carbidopa; Drug: Levodopa/Benzerazide
- Treatment Sequence C (Experimental): Treatment Sequence C Period 1 - 100 mg BIA 9-1067 Period 2 - Placebo Period 3 - 25 mg BIA 9-1067 Period 4 - 50 mg BIA 9-1067
  Levodopa/Carbidopa combination were given to half of the volunteers and Levodopa/Benzerazide to the other half
  Interventions: Drug: BIA 9-1067; Drug: Placebo; Drug: Levodopa/Carbidopa; Drug: Levodopa/Benzerazide
- Treatment Sequence D (Experimental): Treatment Sequence D Period 1 - 50 mg BIA 9-1067 Period 2 - 100 mg BIA 9-1067 Period 3 - Placebo Period 4 - 25 mg BIA 9-1067
  Levodopa/Carbidopa combination were given to half of the volunteers and Levodopa/Benzerazide to the other half
  Interventions: Drug: BIA 9-1067; Drug: Placebo; Drug: Levodopa/Carbidopa; Drug: Levodopa/Benzerazide

INTERVENTIONS:
Drug: BIA 9-1067 — BIA 9-1067 - 25 mg single-dose
  Other Names: OPC, Opicapone
Drug: BIA 9-1067 — BIA 9-1067 - 50 mg single-dose
  Other Names: OPC, Opicapone
Drug: BIA 9-1067 — BIA 9-1067 - 100 mg single-dose
  Other Names: OPC, Opicapone
Drug: Placebo — single-dose
  Other Names: PLC
Drug: Levodopa/Carbidopa — Levodopa 100 mg Carbidopa 25 mg
  Other Names: Sinemet
Drug: Levodopa/Benzerazide — Levodopa 100 mg Benzerazide 25 mg
  Other Names: Madopar®/Restex®

SUMMARY:
The purpose of this study is to investigate the effect of BIA 9-1067 on the levodopa pharmacokinetics when administered in combination with immediate release levodopa/carbidopa or levodopa/benserazide in Parkinson's Disease (PD) patients.

DETAILED DESCRIPTION:
This was a three-centre, double-blind, randomised, placebo-controlled, crossover study with four consecutive single-dose treatment periods in PD patients treated with immediate release 100 mg/25 mg levodopa/carbidopa or 100 mg/25 mg levodopa/benserazide

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-childbearing potential (by reason of surgery or postmenopausal);
* Aged between 30 and 75 years, inclusive;
* A diagnosis of PD according to the UK PDS Brain Bank diagnostic criteria (bradykinesia and at least one of the following: muscular rigidity, rest tremor and postural instability);
* Predictable signs of end-of-dose deterioration despite "optimal" levodopa/carbidopa or levodopa/benserazide therapy;
* Been treated with a stable regimen of 3 to 8 doses of standard release 100 mg/25 mg levodopa/carbidopa or 100 mg/25 mg levodopa/benserazide per day within at least 1 week prior to randomisation;
* Modified Hoehn and Yahr stage of less than 5 in the off-state;
* Mean duration of OFF stage ≥ 1.5 h during waking hours (based on historical information);
* Concomitant anti-Parkinsonian medication (other than apomorphine, entacapone or tolcapone) in stable doses for at least 4 weeks prior to randomisation;
* Results of clinical laboratory tests acceptable by the investigator (not clinically significant for the well-being of the subject or for the purpose of the study);
* Able and willing to give written informed consent.

Exclusion Criteria:

* Non-idiopathic parkinsonism (atypical parkinsonism, symptomatic parkinsonism, Parkinson-plus syndrome);
* Treated with levodopa/carbidopa or levodopa/benserazide in a 10:1 ratio, or with levodopa/carbidopa in a controlled-release formulation;
* Treated with entacapone, tolcapone, neuroleptics, antidepressants (except serotonin-specific reuptake inhibitors or imipramines [desipramine, imipramine, clomipramine and amitriptyline]), monoamine oxidase inhibitors (except selegiline up to 10 mg/day in oral formulation or 1.25 mg/day in buccal absorption formulation or rasagiline up to 1 mg/day) or antiemetics (except domperidone) within 4 weeks prior to randomisation;
* Treated with apomorphine within 7 days prior to randomisation;
* Treated with any investigational product within 2 months prior to randomisation (or within 5 half-lives, whichever is longer);
* A psychiatric or any medical condition that might place him/her at increased risk or interfere with assessments;
* Known hypersensitivity to any of the ingredients of the investigational products;
* A history of abuse of alcohol, drugs or medications within the last 2 years;
* A clinically relevant ECG abnormality;
* A history or current evidence of heart disease, including but not limited to myocardial infarction, angina, congestive heart failure and cardiac arrhythmia;
* Unstable concomitant disease being treated with changing doses of medication;
* A history or current evidence of any relevant disease in the context of this study, i.e., with respect to the safety of the subject (e.g., hepatic or renal impairment) or related to the study conditions;
* A test positive for the human immunodeficiency viruses (HIV) 1 or 2 antibodies, or hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCVAb);
* Donated blood or received blood or blood products within the 6 months prior to randomisation;
* Pregnant, breast-feeding or of childbearing potential;
* Other condition or circumstance that, in the opinion of the investigator, may compromise the subject's ability to comply with the study protocol.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Ferreira, MD, PhD, Principal Investigator — Hospital de Santa Maria, Lisbon
Locations (3):
- Department of Neurology-Hospital de Santa Maria-Faculty of Medicine, University of Lisbon, Lisbon, Portugal
- Spitalul Clinic Colentina - Clinica de Neurologie, Bucharest, Romania
- Department of Neurology- Hospital of the department of medical care of Ministry Internal Affairs of Ukraine, Kyiv, Ukraine

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence A: Period 1 - 25 mg BIA 9-1067 Period 2 - 50 mg BIA 9-1067 Period 3 - 100 mg BIA 9-1067 Period 4 - Placebo
  Levodopa/Carbidopa combination were given to half of the volunteers and Levodopa/Benzerazide to the other half
Period: Overall Study
Arm/Group | Treatment Sequence A | Treatment Sequence B | Treatment Sequence C | Treatment Sequence D
Started | 2 | 2 | 3 | 3
25 mg BIA 9-1067 | 2 | 2 | 3 | 3
50 mg BIA 9-1067 | 2 | 2 | 3 | 3
100 mg BIA 9-1067 | 2 | 2 | 3 | 3
Placebo | 1 | 2 | 3 | 3
Completed | 1 | 2 | 3 | 3
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: The study was to consist of four consecutive treatment periods, corresponding to the 4 different treatment options (25 mg, 50 mg and 100 mg BIA 9-1067or Placebo).According to randomisation, subjects were to receive, in a double-blind manner, 25, 50 and 100 mg BIA 9-1067 or Placebo at 4 separate treatment periods. Each subject were to receive each of the three BIA 9-1067 doses and Placebo in a random sequence with a 3:1 ratio (BIA 9-1067: Placebo) per treatment period.
Arm/Group | Overall Study
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Plasma Concentration Day 3
Description: Cmax - Maximum plasma concentration (ng/mL)
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Placebo: PLC, Placebo
- BIA 9-1067 25 mg; BIA 9-1067 50 mg; BIA 9-1067 100 mg: BIA 9-1067 - OPC, Opicapone
Arm/Group | Placebo | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg
Number analyzed (Participants) | 9 | 10 | 10 | 10
ng/ml
  Cmax (levodopa) | 2103 (48.4) | 2112 (49.6) | 2366 (44.0) | 2657 (32.5)
  Cmax (3-OMD) | 3996 (50.5) | 4193 (42.4) | 4284 (49.2) | 4085 (60.4)
  Cmax (BIA 9-067) | NA (NA) — BIA 9-067 was not administered | 320 (57.2) | 590 (41.5) | 816 (35.5)

2. Secondary Outcome: AUC0-6 - Area Under the Plasma Concentration-time Curve From Time 0 to 6 Hours Post-dose (Day 3)
Description: AUC0-6 - area under the plasma concentration-time curve from time 0 to 6 hours post-dose (ng.h/mL)
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Placebo | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg
Number analyzed (Participants) | 9 | 10 | 10 | 10
ng.h/mL
  AUC0-6 (levodopa) | 3958 (46.7) | 4545 (61.4) | 4580 (36.5) | 5440 (46.4)
  AUC0-6 (3-OMD) | 22334 (51.1) | 22026 (44.3) | 23515 (50.0) | 22200 (61.4)
  AUC0-6 (BIA 9-1067) | NA (NA) — BIA 9-067 was not administered | 776 (60.1) | 1694 (34.6) | 2647 (51.4)

3. Primary Outcome: Tmax = Time to Cmax Day 3
Description: tmax = time to Cmax (values are median)
Time Frame: Day 3
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg
Number analyzed (Participants) | 9 | 10 | 10 | 10
hours
  Tmax (levodopa) | 0.5 [0.5 to 1.5] | 1.0 [0.5 to 2.0] | 0.5 [0.5 to 2.0] | 0.5 [0.5 to 1.5]
  Tmax (3-OMD) | 2.00 [0.0 to 3.0] | 1.75 [0.0 to 4.0] | 2.50 [0.0 to 4.0] | 1.75 [1.0 to 6.0]
  Tmax (BIA 9-067) | NA [NA to NA] — BIA 9-067 was not administered | 2.00 [0.5 to 3.0] | 2.00 [1.0 to 6.0] | 2.00 [1.0 to 4.0]

ADVERSE EVENTS:
Time Frame: 10 months
Groups:
- 25 mg BIA 9-1067: 25 mg BIA 9-1067 ESL, Eslicarbazepine
- 50 mg BIA 9-1067: 50 mg BIA 9-1067 ESL, Eslicarbazepine
- 100 mg BIA 9-1067: 100 mg BIA 9-1067 ESL, Eslicarbazepine
- Placebo: Placebo ESL, Eslicarbazepine
Arm/Group | 25 mg BIA 9-1067 | 50 mg BIA 9-1067 | 100 mg BIA 9-1067 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 5/10 | 6/10 | 7/10 | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 25 mg BIA 9-1067 (N=10) | 50 mg BIA 9-1067 (N=10) | 100 mg BIA 9-1067 (N=10) | Placebo (N=9)
EOSINOPHIL PERCENTAGE INCREASED (Investigations) | 0 | 1 | 1 | 1
TACHYCARDIA (Cardiac disorders) | 0 | 1 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
SOMNOLENCE (Nervous system disorders) | 0 | 1 | 1 | 1
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 | 0 | 1 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 1 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 1
PALLOR (Vascular disorders) | 0 | 0 | 0 | 1
RESPIRATORY INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 1 | 1 | 0
HALLUCINATION (Psychiatric disorders) | 0 | 0 | 0 | 1
BLOOD PRESSURE INCREASED (Investigations) | 0 | 1 | 0 | 0
LIGHTHEADEDNESS (Nervous system disorders) | 0 | 1 | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 1 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0
HYPOTENSION (Vascular disorders) | 0 | 1 | 0 | 0
INSOMNIA (Psychiatric disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other